CLINICAL TRIAL: NCT05705050
Title: Effect of Intraoperative Aminophylline Infusion on Pain Intensity After Ureterocopic Lithotripsy Surgeries
Brief Title: Aminophylline Infusion on Pain Intensity After Ureterocopic Lithotripsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Osama Rehab, Lecturer of Anesthesiology, Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR19/1/23
Record Dates: First submitted 2023-01-21; First posted 2023-01-30 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Aminophylline; Pain; Ureterocopic Lithotripsy
Keywords: Aminophylline; Postoperative Pain; Ureterocopic Lithotripsy
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aminophylline group (Experimental): Patients will receive 4 mg/kg aminophylline diluted in 100 ml normal saline over 20 minutes after induction of anesthesia and positioning of patients in lithotomy position.
  Interventions: Drug: Aminophylline group
- Control group (Placebo Comparator): Patients will receive 100 ml normal saline over 20 minutes after induction and lithotomy positioning.
  Interventions: Other: Control group

INTERVENTIONS:
Drug: Aminophylline group — Patients will receive 4 mg/kg aminophylline diluted in 100 ml normal saline over 20 minutes after induction of anesthesia and positioning of patients in lithotomy position.
  Arms: Aminophylline group
Other: Control group — Patients will receive 100 ml normal saline over 20 minutes after induction and lithotomy positioning.
  Arms: Control group

SUMMARY:
This study will be conducted to evaluate the effect of intraoperative systemic aminophylline infusion on pain intensity in patients undergoing ureteroscopic lithotripsy surgeries with ureteric stent placement at the end of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 to 50 years
* American society of anesthesiology (ASA) physical status I - II
* Body mass index (BMI) less than 30.0 kg/m2
* Scheduled for ureteroscopic lithotripsy surgery with D-J ureteric stent placement at the end of procedure
* Under general anesthesia.

Exclusion Criteria:

1. Patients with central nervous system diseases, cardiovascular diseases, arrhythmias, cerebrovascular diseases, convulsions, renal impairment or hepatic dysfunction.
2. Pregnancy or lactation.
3. Patients with a history of allergy to aminophylline.
4. Coffee consumption (more than 2 cups/day)
5. Patients with opioid addiction or patients treated with B agonists, tranquilizers, or antidepressants.
6. Short procedures less than 30 minutes or procedures not requiring D-J stent placement.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-06-18 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Intensity of pain | In post anesthesia care unit (PACU)
  Visual analogue score (VAS) score: will be measured on arrival to PACU, at 30 minutes, 1 hour, 2 hour, 6, 12 and 24 hour after surgery.

SECONDARY OUTCOMES:
Intensity of pain | 24 hour after surgery
  Visual analogue score (VAS) score: will be measured on arrival to PACU, at 30 minutes, 1 hour, 2 hour, 6, 12 and 24 hour after surgery.
Total amount of opioid dose | 24 hour after surgery
  If Patients reported VAS score more than 3, they will receive intravenous 0.5 mg /kg pethidine. All patients will be observed in PACU for at least 2 hour and in the ward on the day of surgery for confirming any side effects or complications.
The incidence of postoperative adverse reactions | 24 hour after surgery
  the incidence of adverse reactions, such as arrhythmia, postoperative nausea and vomiting (PONV) and postoperative lightheadedness will be recorded in both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, ElGharbiaa, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available 6 months after publication
Access Criteria: The data will be available upon a reasonable request from the corresponding author